CLINICAL TRIAL: NCT01738152
Title: A Single-Arm Clinical Trial Investigating the Feasibility of a Non-Hormonal Vaginal Moisturizer in Hormone-Receptor Positive Postmenopausal Cancer Survivors Experiencing Estrogen Deprivation Symptoms on Vulvovaginal Health
Brief Title: Non-Hormonal Vaginal Moisturizer in Hormone-Receptor Positive Postmenopausal Cancer Survivors Experiencing Estrogen Deprivation Symptoms on Vulvovaginal Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-232
Record Dates: First submitted 2012-11-28; First posted 2012-11-30 (Estimated); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Breast Cancer; Endometrial Cancer
Keywords: HYALOGYN VAGINAL GEL; vaginal dryness; 12-232
MeSH Terms: conditions — Breast Neoplasms; Endometrial Neoplasms | interventions — Surveys and Questionnaires

ARMS (1):
- HLA treatment (Experimental): This is a single arm prospective longitudinal clinical trial investigating the feasibility of a hyaluronic acid (HLA) vaginal gel (HyaloGYN®; Cebert Pharmaceuticals, Inc.; Birmingham, Alabama) to improve estrogen deprivation vaginal and vulvar health symptoms in post-menopausal women with a history of hormone-receptor positive cancer with estrogen deprivation symptoms of vaginal dryness and discomfort.
  Interventions: Other: HLA vaginal gel (HyaloGYN®),; Behavioral: questionnaires

INTERVENTIONS:
Other: HLA vaginal gel (HyaloGYN®), — Each participant will receive a HLA vaginal gel (HyaloGYN®), which is an over-the-counter, colorless gel to be administered for hydration and lubrication of the vaginal epithelium for women suffering dryness,as well as to the vulva for women suffering from vulvar symptoms. All participants will be instructed to insert the HLA gel into the vagina (with applicator) daily for the first 2 weeks, and then 3 times per week for 10 weeks. The women with vulvar symptoms at the baseline assessment will additionally be instructed to apply the HLA gel onto the vulva (manually) daily for the first 2 weeks, and then 3 times per week for 10 weeks. The participants will be assessed at 12 weeks. Participants receiving benefit from HyaloGYN®, as operationalized by improvement in both vaginal pH and VAS score will continue using the product 3 times per week for another 12 weeks and will receive a final vulvovaginal assessment at 24 weeks post-HLA treatment initiation.
Behavioral: questionnaires — Assessment Form as part of routine clinical care. Participants will be asked to complete questionnaires at the baseline initial evaluation, 4-6 weeks, 12-14 weeks, and 22-24 weeks. The study information collected will be found in the standardized Clinical Assessment Form that patients complete as part of routine clinical care, along with an additional survey pertinent to the aims of the study. At 24 weeks, participants will complete an additional questionnaire that will ask questions regarding their experience with HyaloGYN® and their acceptability of and satisfaction with the product. Study participants must see the FSM NP or GYN clinician for the targeted exams at the study follow-up time points (4-6 weeks, 12-14 weeks, 22-24 weeks). PhD follow-up visits can be based upon the treatment plan of the patient. The study questionnaires and moisturizer diaries will be completed and collected during follow-up appointments with the GYN clinician or FSM NP.

SUMMARY:
The purpose of this study is to see whether it is feasible to conduct a study to determine if the use of hyaluronic acid (HLA) vaginal gel (HyaloGYN®) improves vulvovaginal health.

This study aims to look at whether or not HyaloGYN® is effective in women with a history of hormone receptor positive cancer and experiencing vaginal and/or vulvar symptoms of estrogen deprivation following their breast and endometrial cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* History of breast cancer or endometrial cancer confirmed at MSKCC or outside pathology report
* Breast cancer patients must be at least 3 months post-active treatment (including chemotherapy, radiation therapy, endocrine therapy, and/or maintenance therapy), but not greater than 5 years post-active treatment (exception: AIs are required, and monoclonal antibodies are allowed)
* Breast cancer patients must be currently on adjuvant aromatase inhibitors
* Endometrial cancer patients must be at least 3 months post-active chemotherapy and/or maintenance therapy treatment but not greater than 5 years post-active chemotherapy and/or maintenance therapy treatment. They must be at least 4 weeks post-radiation therapy (EBRT or IVRT) but not greater than 5 years post-radiation therapy.
* Endometrial cancer patients must have underwent surgical treatment (total abdominal hysterectomy ([TAH]/BSO)) and radiation therapy (external beam radiation therapy [EBRT] or IVRT)
* Currently have no clinical evidence of disease
* Menopausal at study entry as described by:
* Surgical menopause (TAH/BSO), or
* Age ≥ 50 years and cessation of menstruation for at least 1 year, or
* Age <50 years and cessation of menstruation for at least 1 year with estradiol level in post-menopausal range, or
* Rendered post-menopausal with the use of LHRH agonist
* Patients who are new visits to Female Sexual Medicine Program or patients are not consistently using any vulvovaginal health promotion strategies (e.g., pelvic floor exercises, dilator therapy, moisturizers) recommended by the Female Sexual Medicine Program Reporting being bothered by vulvovaginal symptoms of estrogen deprivation (i.e., vulvovaginal dryness or discomfort [pain with intercourse or examination])
* Without history of other cancers (excluding non-melanoma skin cancer)
* Women at least 18 years of age
* Able to read and speak English
* Able to participate in the informed consent process

Exclusion Criteria:

* Inability to provide informed consent
* Vaginal bleeding of unknown etiology within 12 months of study entry
* Currently taking hormone replacement therapy [local or systemic] (Patients must discontinue for 2 weeks in order to be eligible prior to study enrollment)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2012-11; Primary Completion 2021-07-21 (Actual); Study Completion 2021-07-21 (Actual)

PRIMARY OUTCOMES:
investigate feasibility of conducting a 12-week HLA treatment regimen | 12-week
  a 12-week HLA treatment regimen, as defined by the percentage of women who are evaluable at the 12-week assessment (i.e., women who have completed both baseline and 12-week vaginal and vulvar outcome assessments).

SECONDARY OUTCOMES:
Vaginal Assessment Composite Score [VAS] | 12 weeks post-HLA treatment initiation
  as measured by the Vaginal Assessment Composite Score [VAS], vaginal pH and epithelial atrophy)
Vulvar Assessment Composite Score [VuAS] | 12 weeks post-HLA treatment initiation
  (as measured by the Vulvar Assessment Composite Score [VuAS], vulvar atrophy, and vulvar/vestibular irritation)

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne Carter, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/